CLINICAL TRIAL: NCT06494098
Title: Conventional Versus Modified Pre-surgical Naso-Alveolar Molding Treatment in Cleft Lip and Palate Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02204023PP
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2023-09

CONDITIONS: Cleft Lip and/or Palate; Cleft Lip Bilateral
Keywords: Cleft palate; Cleft Lip and/or Palate; Nasoalveolar Molding
MeSH Terms: conditions — Cleft Palate | interventions — Nasoalveolar Molding

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAM group (Experimental)
  Interventions: Procedure: Nasoalveolar Molding; Diagnostic Test: Addition silicone impression
- MNAM (Experimental)
  Interventions: Procedure: Nasoalveolar Molding; Diagnostic Test: Addition silicone impression

INTERVENTIONS:
Procedure: Nasoalveolar Molding — presurgical orthopedics
Diagnostic Test: Addition silicone impression — diagnostic impression for maxillary arch and nose

SUMMARY:
The aim of this study is to evaluate and compare clinically conventional Pre-surgical Naso-Alveolar Molding (PNAM) treatment versus Modified Naso-Alveolar Molding protocol (MPNAM) in cleft lip and palate patients in terms of:

1. Decreasing cleft gap.
2. Attaining columellar length.
3. Effect on maxillary growth.
4. Treatment Duration.
5. Parents acceptance.

ELIGIBILITY:
Inclusion Criteria:

1. The age range from 14 -30 days after birth.
2. Has complete cleft lip and palate.
3. Parents acceptance.
4. Medically free infants.

Exclusion Criteria:

1. Syndromic patients.
2. Medically compromised patients contradicting operation.

Ages: 2 Weeks to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-06-16 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Attaining columellar length | 3 month
  the length of columella has increased after nasoalveolar molding orthopedic treatment

SECONDARY OUTCOMES:
Treatment Duration | 3 month
  the time taken to decrease the alveolar cleft gap and to lengthen the columella

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://mjd.journals.ekb.eg/article_223404_d6468537a8523931419282df147cbe16.pdf